CLINICAL TRIAL: NCT05497492
Title: Comparison of the Effects of Esketamine, Sufentanil, or Lidocaine Combined With Propofol on Tussis Reflection During Upper Gastroscopy: a Randomised, Two Centre, Three-blind, Controlled Trial
Brief Title: Comparison of the Effects of Esketamine, Sufentanil, or Lidocaine on Tussis Reflection During Upper Gastroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: lumen208
Record Dates: First submitted 2022-07-19; First posted 2022-08-11 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia
Keywords: gastroscopy; esketamine; sufentanil; lidocaine; propofol; tussis
MeSH Terms: interventions — Propofol; Sufentanil; Esketamine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- P group (Active Comparator): single administration of propofol
  Interventions: Drug: propofol
- P + S group (Experimental): administration of propofol and sufentanil in combination
  Interventions: Drug: propofol and sufentanil
- P + K group (Experimental): administration of propofol and esketamine in combination
  Interventions: Drug: propofol and esketamine
- P + L group (Experimental): administration of propofol and lidocaine in combination
  Interventions: Drug: propofol and lidocaine

INTERVENTIONS:
Drug: propofol — single administration of propofol
  Other Names: P
  Arms: P group
Drug: propofol and sufentanil — administration of propofol and sufentanil in combination
  Other Names: P+S
  Arms: P + S group
Drug: propofol and esketamine — administration of propofol and esketamine in combination
  Other Names: P+K
  Arms: P + K group
Drug: propofol and lidocaine — administration of propofol and lidocaine in combination
  Other Names: P+L
  Arms: P + L group

SUMMARY:
the frequency of tussis, nausea and vomiting, and/or body movements observed at the insertion of the endoscope into the pharyngeal cavity or within 5 min of endoscope insertion.

DETAILED DESCRIPTION:
The patients are selected according to their inclusion and exclusion criteria for diagnostic upper GI endoscopy and informed consent. The patients will be divided into the four groups: P group (single administration of propofol), P + S group (administration of propofol and sufentanil in combination), P + K group (administration of propofol and esketamine in combination), and P + L group (administration of propofol and lidocaine in combination) (N = 100 per group). Baseline information will be collected and recorded before the operation. Anaesthetic drugs will be prepared by the nurses and anaesthetists on the day of the operation as follows: 0.9% normal saline (20 mL) for the P group, 0.5 μg/mL sufentanil (20 mL) for the P + S group, 1.5 mg/mL esketamine (20 mL) for the P + K group, and 10 mg/mL lidocaine (20 mL) for the P + L group. Before entering the operating room, the patients will be given lidocaine defoamer for gargling to open the upper limb vein and 5 mL/min Lactate Ringer solution. After entering the room, the patients will wear masks to inhale high-flow oxygen, and their vital signs will be monitored and recorded as Tire. Analgesic drugs (diluted to 20 mL according to different concentrations) prepared by the nurses will be slowly injected into their veins 5 min before examination for 30 s (the dose was calculated using the formula: the injected drug dose (ml) = the weight of the patient (kg)/10"; 1.5 mg/kg propofol will be intravenously administrated. . Multiple-dose administration is acceptable according to the state of the patient. The endoscope will be inserted when the eyelash reflex disappeared (sedation depth grade: deep sedation). Blood pressure will be recorded after every 3 min from the beginning of the examination, and HR, SpO2, and RR will be recorded simultaneously. The frequency and degree of tussis, nausea, and vomiting and/or body movements at endoscope insertion or within 5 min of insertion will be monitored. In case of any abnormalities, they should be described in detail, and appropriate doses of propofol should be added until the endoscope exits the teeth pad. During endoscopy, 2-4 mL of propofol should be added under the conditions of extended operation time, accelerated breathing, and elevated blood pressure and heart rate to maintain deep sedation. The patients will be transferred to a recovery room after the operation, and their vital signs will be recorded after every 5 min until the patients met the standard of leaving the hospital (Steward score ≥ 4) before discharge

ELIGIBILITY:
Inclusion Criteria

* undergoing diagnostic upper GI endoscopy under deep propofol sedation
* >18 year old
* meeting the classification I-III of American Society of Anesthesiologists (ASA)
* getting written informed consent

Exclusion Criteria:

* allergic reaction to planned medication
* gravis myasthenia
* history of psychological problems or psychiatric disease
* morbid obesity/obstructive sleep apnea
* acute upper respiratory infections
* asthma at acute stage
* history of unregulated or malignant hypertension
* history of significant ischemic heart disease or severe arrhythmia
* severe liver or kidney dysfunction or coagulation disorders
* acute upper GI haemorrhage with shock
* severe anaemia
* GI obstruction with gastric retention
* seizure disorders
* long-term history of sedative and analgesic drug use
* increased intracranial pressure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
the frequency of tussis, nausea and vomiting, and/or body movements observed at the insertion of the endoscope into the pharyngeal cavity or within 5 minutes of endoscope insertion. | an average of 5 minutes，at the insertion of the endoscope into the pharyngeal cavity or within 5 minutes of endoscope insertion
  the frequency of tussis

SECONDARY OUTCOMES:
recovery time | an average of 30 minutes，the time from withdrawal of endoscopy to obeying verbal commands
  recovery time from anesthesia
propofol dosage during operation | through study completion, an average of 20 minutes，the time from insertion endoscopy to withdrawal of endoscopy
  propofol dosage during operation
incidence of perioperative adverse events | through study completion, an average of 1 year，the time from insertion endoscopy to withdrawal of endoscopy
  incidence of perioperative adverse events
incidence of postoperative adverse events | through study completion, an average of 1 year，
  incidence of postoperative adverse events
MMSE scores after operation | through study completion, an average of 1 year after operation
  MMSE scores

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Hou, MD, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Triantafillidis JK, Merikas E, Nikolakis D, Papalois AE. Sedation in gastrointestinal endoscopy: current issues. World J Gastroenterol. 2013 Jan 28;19(4):463-81. doi: 10.3748/wjg.v19.i4.463. PMID 23382625
- [Result] Canning BJ. Afferent nerves regulating the cough reflex: mechanisms and mediators of cough in disease. Otolaryngol Clin North Am. 2010 Feb;43(1):15-25, vii. doi: 10.1016/j.otc.2009.11.012. PMID 20172253
- [Result] Wehrmann T, Triantafyllou K. Propofol sedation in gastrointestinal endoscopy: a gastroenterologist's perspective. Digestion. 2010;82(2):106-9. doi: 10.1159/000285554. Epub 2010 Apr 21. PMID 20407257
- [Result] Byrne MF, Chiba N, Singh H, Sadowski DC; Clinical Affairs Committee of the Canadian Association of Gastroenterology. Propofol use for sedation during endoscopy in adults: a Canadian Association of Gastroenterology position statement. Can J Gastroenterol. 2008 May;22(5):457-9. doi: 10.1155/2008/268320. PMID 18478130
- [Result] Ho WM, Yen CM, Lan CH, Lin CY, Yong SB, Hwang KL, Chou MC. Comparison between the recovery time of alfentanil and fentanyl in balanced propofol sedation for gastrointestinal and colonoscopy: a prospective, randomized study. BMC Gastroenterol. 2012 Nov 21;12:164. doi: 10.1186/1471-230X-12-164. PMID 23170921
- [Result] Poulos JE, Kalogerinis PT, Caudle JN. Propofol compared with combination propofol or midazolam/fentanyl for endoscopy in a community setting. AANA J. 2013 Feb;81(1):31-6. PMID 23513321
- [Result] Zhang L, Bao Y, Shi D. Comparing the pain of propofol via different combinations of fentanyl, sufentanil or remifentanil in gastrointestinal endoscopy. Acta Cir Bras. 2014 Oct;29(10):675-80. doi: 10.1590/s0102-8650201400160008. PMID 25318000
- [Derived] Hou HJ, Liu L, Tian M, Xue FS. Comparison of the effects of esketamine, sufentanil, or lidocaine combined with propofol on tussis reflection during upper gastrointestinal endoscopy: study protocol for a randomised, two centre, three-blind, controlled trial. Trials. 2024 Jan 4;25(1):24. doi: 10.1186/s13063-023-07812-0. PMID 38178168